CLINICAL TRIAL: NCT04062461
Title: A Multicenter Randomized Clinical Trial Aimed at Evaluating the Effectiveness of Self-care Promotion in Patients With Heart Failure
Brief Title: Evaluate the Effectiveness of Self-care Multifaceted Strategy in Heart Failure Patients
Acronym: IC-CBC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital do Coracao (Other)
Collaborators: Hospital Moinhos de Vento (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2019-06-13; First posted 2019-08-20 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: A randomized, multicenter, national, phase II clinical trial aimed at evaluating the effectiveness of self-care promotion using a multifaceted strategy based on sending text messages SMS to patients with heart failure.
Who Masked: Outcomes Assessor
Masking Description: Experimental group:
  -Self-care promotion using a multifaceted strategy based on the use of a tele-monitoring device, based on short message system (SMS) messages and self-care teaching tools.
  Patients will receive daily messages to optimize self-care in heart failure with the following functions:
  * customized reminders about medication schedules
  * weight and symptoms of decompensation monitoring assessing a decision tree with diuretics adjustment if needed and alerts that define the need to contact a health professional for early intervention before deterioration of the clinical state, identifying situations that require clinical intervention.
  * educational content on heart failure for the patient (symptoms of the disease, healthy habits for HF, warning signs for severity)
  * diary for registration of visits to health services and clinical setting.
  Control group:
  -Usual outpatient care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-care promotion (Experimental): multifaceted strategy based on sending text messages(SMS) to patients with heart failure.
  Press educational content on heart failure for the patient (symptoms of the disease, healthy habits for HF, warning signs for severity).
  The text messages are about how the patient should take your drugs (evem diuretics), measure blood pressure and weight in Kg, and about signals and symptoms (shorthbreathness during the night), and about how important is practice physical exercises and don't drink alcohol.
  Interventions: Other: Multifaceted strategy based on sending text messages(SMS)
- Control group (Active Comparator): routinely management in the HF. Press educational content on heart failure for the patient (symptoms of the disease, healthy habits for HF, warning signs for severity)
  Interventions: Other: Usual outpatient care

INTERVENTIONS:
Other: Multifaceted strategy based on sending text messages(SMS) — multifaceted strategy based on sending text messages(SMS) to patients with heart failure.
  Press educational content on heart failure for the patient (symptoms of the disease, healthy habits for HF, warning signs for severity).
  The text messages are about how the patient should take your drugs (evem diuretics), measure blood pressure and weight in Kg, and about signals and symptoms (shorthbreathness during the night), and about how important is practice physical exercises and don't drink alcohol.
  Arms: self-care promotion
Other: Usual outpatient care — Educational content on heart failure for the patient (symptoms of the disease, healthy habits for HF, warning signs for severity)
  Arms: Control group

SUMMARY:
Study Design: A randomized, multicenter, national, phase II clinical trial aimed at evaluating the effectiveness of self-care promotion using a multifaceted strategy based on sending text messages(SMS)to patients with heart failure.

Methodological quality:

* Central randomization with allocation concealment;
* Decision committee for blind outcome assessment;
* Intention-to-treat analysis

DETAILED DESCRIPTION:
Study Design -A randomized, multicenter, national, phase II clinical trial aimed at evaluating the effectiveness of self-care promotion using a multifaceted strategy based on sending text messages(SMS) to patients with heart failure.

Methodological quality

-Central randomization with allocation concealment; Decision committee for blind outcome assessment; Intention-to-treat analysis

Primary Objective -To develop and evaluate the feasibility of a monitoring, education and self-care strategy to optimize the management of patients with heart failure (HF) after hospital discharge.

Secondary Objectives

-To evaluate, in patients with heart failure, the effect of a self-care promotion program using a multifaceted strategy in comparison to the usual care about acceptability to the application of SMS, patient and / or family satisfaction with care, quality of life scales health scales, self-care scales and knowledge on HF, visual analog scale of dyspnea, and clinical outcomes at 30 and 180 days.

Experimental group:

-Self-care promotion using a multifaceted strategy based on the use of a tele-monitoring device, based on short message system (SMS) messages and self-care teaching tools.

Patients will receive daily messages to optimize self-care in heart failure with the following functions:

* customized reminders about medication schedules
* weight and symptoms of decompensation monitoring assessing a decision tree with diuretics adjustment if needed and alerts that define the need to contact a health professional for early intervention before deterioration of the clinical state, identifying situations that require clinical intervention.
* educational content on heart failure for the patient (symptoms of the disease, healthy habits for HF, warning signs for severity)
* diary for registration of visits to health services and clinical setting.

Control group:

-Usual outpatient care

Follow-up

* Follow up will be at least 180 days from the inclusion in the study.
* Sample size estimation 350 patients per group (700 patients)

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years)
* Heart failure of any etiology
* Vulnerable period after episode of acute decompensation
* Cellular telephony acess;
* Left Ventricular Ejection Fraction (LVEF <40%),

Exclusion Criteria:

* Cardiac transplant wait list;
* Surgical or percutaneous (coronary or valvular) treatment at last 3 months
* HF terminal ;
* Life expectancy <1 year;
* Another drug or device study at last 30 days
* Prior randomization in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
The evaluation of the effect of multifaceted intervention compared to usual outpatient care on the primary endpoint will be performed using the Student's t-Student test of the log ratio of NT-proBNP levels at 6 months baseline. | six months
  Variation of NT-proBNP in 180 days;

SECONDARY OUTCOMES:
Overall mortality | Six months
  Overall mortality for Heart Failure at 180 days
Overall hospitalization | Six months
  Overall hospitalization for Heart Failure at 180 days
Cardiovascular mortality | Six months
  To evaluate cardiovascular mortality in 180 days
Emergency department visit | Six months
  To evaluate emergency department visit in 180 days
Satisfaction of the patient and / or caregiver with health care | Thirty days
  Using (NPS tool):Scale of 0-10 to measure satisfaction of the patient and / or caregiver with health care. Rate it from 0 to 10, where 0 means not at all satisfied and 10 means extremely satisfied.
Acceptability / adherence to the system of sending messages | Six months
  Using a Scale of 0-10 (question to insert the note) to measure acceptability / adherence to the system of sending messages. Rate it from 0 to 10, where 0 means no help at all and 10 means the posts were extremely beneficial.
Variation of NT-proBNP in 30 days | 30 days
  The evaluation of the effect of multifaceted intervention compared to usual outpatient care on the primary endpoint will be performed using the Student's t-Student test of the log ratio of NT-proBNP levels at 30 days from baseline.
Kansas Health-related quality of life in baseline, 30 and 180 days | From baseline, 30 and 180 days.
  Using (Kansas Health-related quality of life Questionnaire): Scale of 0-100 to measure quality of life in patients with heart failure. Rate it from 0 to 100. Overall score means higher is better.
Variation scale numeric of VAS (Visual Analogue Scale) of dyspnea. | Baseline, 30, 90 and 180 days visits
  Using Variation scale numeric of VAS (Visual Analogue Scale) to measure degree of dyspnea. Rate from 0 to 10, where 0 means no dyspnea and 10 the highest complain of dyspnea.
European Heart Failure Self-Care Behavior Scale - EHFScBs | From 30 and 180 days.
  Using (EHFScBs): Scale of 0-60 to to measure self-care behavior of heart failure (HF) patients. Rate it from 0 to 60. Overall score means smaller is better.
Heart Failure Knowledge Questionnaire | From 30 and 180 days.
  Used to measure Knowledge about Heart Failure. Are by 14 questions more than 70% of correct answers means good Knowledge.

OTHER OUTCOMES:
Win Ratio Analysis | 6 months
  A pre-specified analysis using the win ratio method will be performed. A composite outcome will be analysed in the hierarchical order of 1) time to cardiovascular death; 2) time to first hospitalization due to heart failure; 3) relative change in NT-proBNP from baseline to 180 days. In this last comparison, to have a winner, the relative change needs to differ by more than 20% between two subjects. By the protocol, all the clinical outcomes (including CV death and HF hospitalization) will be assessed until 6 months.
Subgroup Analysis | Variables at baseline and primary outcome at 6 months
  Analysis of the primary endpoint will be performed in pre-specified subgroups: age strata, gender, educational levels, New York Heart Association functional classes, left ventricular ejection fraction strata, NT-proBNP levels, HF aetiology, baseline KCCQ scores, and baseline HF self-care and knowledge scores.
Analysis according to renal function | Renal function at baseline and study endpoints at 6 months
  Analysis of study endpoints (cardiovascular mortality, hospitalization due to heart failure and NT-proBNP variation) will be performed according to baseline renal function strata.

CONTACTS AND LOCATIONS:
Overall Officials: Félix J Alvarez Ramires, Alvarez Ramires, Principal Investigator — Hospital do Coração - HCor; Luiz E Rohde, MD,PhD, Principal Investigator — Hospital Moinhos de Vento
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rohde LE, Rover MM, Hoffmann Filho CR, Rabelo-Silva ER, Silvestre OM, Martins SM, Passos LCS, de Figueiredo Neto JA, Danzmann LC, Silveira FS, Mesas CE, Hernandes ME, Moura LZ, Simoes MV, Ritt LEF, Nishijuka FA, Bertoldi EG, Dall Orto FTC, Magedanz EH, Mourilhe-Rocha R, Fernandes-Silva MM, Ferraz AS, Schwartzmann P, de Castilho FM, Pereira Barretto AC, Dos Santos Junior EG, Nogueira PR, Canesin M, Beck-da-Silva L, de Carvalho Silva M, Adolfi Junior MS, Santos RHN, Ferreira A, Pereira D, Lopez Pedraza L, Kojima FCS, Campos V, de Barros E Silva PGM, Blacher M, Cavalcanti AB, Ramires F; MESSAGE-HF Investigators. Multifaceted Strategy Based on Automated Text Messaging After a Recent Heart Failure Admission: The MESSAGE-HF Randomized Clinical Trial. JAMA Cardiol. 2024 Feb 1;9(2):105-113. doi: 10.1001/jamacardio.2023.4501. PMID 38055237
- [Derived] Rohde LE, Hoffmann Filho CR, Rover MM, Rabelo-Silva ER, Lopez L, Passos LCS, Silvestre OM, Martins SM, de Figueiredo Neto JA, Silveira FS, Canesin MF, Simoes MV, Akio Nishijuka F, Bertoldi EG, Danzmann LC, Mourilhe-Rocha R, Magedanz EH, Esteves M, de Castilho FM, Fernandes-Silva MM, Ritt LEF, Blacher M, Soares RM, Cavalcanti AB, Ramirez F. Design of a multifaceted strategy based on automated text messaging in patients with recent heart failure admission. ESC Heart Fail. 2021 Dec;8(6):5523-5530. doi: 10.1002/ehf2.13516. Epub 2021 Sep 18. PMID 34535979